CLINICAL TRIAL: NCT05731401
Title: Expressed Beliefs About the Cause of Pain in a Paediatric Population: a Mixed Explanatory Sequential Study.
Brief Title: Expressed Beliefs About the Cause of Pain in a Paediatric Population
Acronym: EBPain
Status: Completed | Type: Observational
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Laura Menés Fernández, Principal Investigator, University Rovira i Virgili
Other Study IDs: 114/2018
Record Dates: First submitted 2023-01-24; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Chronic Pain; Pediatric ALL; Pain Perception
MeSH Terms: conditions — Chronic Pain; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Explanations of the cause of pain — When analyzing the responses to the question "Why do you think you have or have had this pain?" two themes emerged from the data: 'explanations associated with damage', and 'explanations not associated with damage'.
  The themes were sub-classified into sub-themes, according to the type of explanation

SUMMARY:
The aims of this study are to explore what beliefs children and adolescents manifest about the cause of the pain they describe; to compare whether if there are differences between beliefs by age and by persistence of pain; and to relate explanations of the cause of pain with current scientific evidence to determine if these beliefs are erroneous.

DETAILED DESCRIPTION:
Design:

Mixed (explanatory sequential). The primary endpoint of the study were explanations of the cause of pain recorded by means of an open-ended question.

Setting:

The participants were school-age children attending a charted school in the province of Barcelona.

Participants:

Of the 345 potential school participants, 306 agreed to participate. 36 pupils were excluded when applying the eligibility criteria, so the resulting sample was of 270.

ELIGIBILITY:
Inclusion Criteria:

* to be schooled at the El Cim school
* to be between 10 and 16 years old (both included)
* to have or have had pain in the last month; to be able to read and write in Catalan and/or Spanish.

Exclusion Criteria:

* had an intellectual disability and/or cognitive impairment that interfered with their participation
* had not submitted the informed consent form duly completed and signed by their legal guardians

Ages: 10 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: The participants in this study were a convenience sample of schoolchildren aged 10- 16 years from a charter school (Barcelona, Spain), a school large enough to have a sufficient sample.
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Explanations of the cause of pain | 1 year
  Participants were asked to fill out a questionnaire where they were asked "Do you have or have you had pain in the last month?" and "Why do you think you have or have had this pain?".
  The answer is an open response.

CONTACTS AND LOCATIONS:
Locations (1):
- Laura Menés Fernández, Vilanova i la Geltrú, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pate JW, Noblet T, Hush JM, Hancock MJ, Sandells R, Pounder M, Pacey V. Exploring the concept of pain of Australian children with and without pain: qualitative study. BMJ Open. 2019 Oct 28;9(10):e033199. doi: 10.1136/bmjopen-2019-033199. PMID 31662406
- [Background] Salvat I, Adillon C, Andres EM, Monterde S, Miro J. Development of the Conceptualization of Pain Questionnaire: A Measure to Study How Children Conceptualize Pain. Int J Environ Res Public Health. 2021 Apr 6;18(7):3821. doi: 10.3390/ijerph18073821. PMID 33917429
- [Background] Huguet A, Miro J. The severity of chronic pediatric pain: an epidemiological study. J Pain. 2008 Mar;9(3):226-36. doi: 10.1016/j.jpain.2007.10.015. Epub 2007 Dec 21. PMID 18088558
- [Background] Hassett AL, Hilliard PE, Goesling J, Clauw DJ, Harte SE, Brummett CM. Reports of chronic pain in childhood and adolescence among patients at a tertiary care pain clinic. J Pain. 2013 Nov;14(11):1390-7. doi: 10.1016/j.jpain.2013.06.010. Epub 2013 Sep 7. PMID 24021576